CLINICAL TRIAL: NCT05497427
Title: Normative Database and Test-Retest Reliability for BrainCheck Assessments
Acronym: NDTR
Status: Completed | Type: Observational
Sponsor: BrainCheck, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00064230
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change; Cognitive Decline; Cognitive Deterioration; Neurocognitive Deficit
Keywords: Healthy Volunteers; Dementia; Alzheimer's Disease; Mild Cognitive Impairment; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Normative: BrainCheck assessment values from participants that have indications of healthy cognition at the time of testing ( a SLUMS result considered 'normal', more than 4 hours of sleep the night before, not having consumed alcohol or drugs within the last 6 hours, or not have participated in high capacity and strenuous physical activity within the last hour.)
  Interventions: Device: BrainCheck Assessment
- Test-Retest: Comparing BrainCheck assessment values between an initial visit test and a follow-up visit test 7-14 days later within subjects.
  Interventions: Device: BrainCheck Assessment
- Per Protocol: BrainCheck assessment values from participants that completed all procedures with no protocol deviations
  Interventions: Device: BrainCheck Assessment

INTERVENTIONS:
Device: BrainCheck Assessment — A computerized neurocognitive test administered via an electronic device, such as a phone, tablet or computer, that contains several assessments that will aid in establishing an individuals cognitive performance

SUMMARY:
The purpose of this study is to collect normative test values and demographic information for normative and referential data for a rapid, portable, computerized neurocognitive testing device from healthy adults 50 and older.

DETAILED DESCRIPTION:
BrainCheck's battery of 12 cognitive assessments will be used in this study, which aims to measure a variety of cognitive domains (memory, attention, mental flexibility, executive function, processing speed, balance, reasoning, visuospatial construction, language, and visual hallucinations).

With the decline in cognition occurring at a quicker rate at older ages, this study aims to collect additional data from healthy older adults to better capture the normative distribution among these age groups from existing and new assessments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or older
* Willing and able to comply with study requirements and activities

Exclusion Criteria:

* TBI within the last 6 months
* Neurosurgery within the last month
* Experienced a stroke
* Self reported neurological condition (including mild neuropsychological impairment, dementia, Parkinson's disease, amyotrophic lateral sclerosis, Multiple sclerosis, or long-covid)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy volunteers 50 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Mean, standard deviation, and percentiles of values of BrainCheck Assessments | 5 months
  BrainCheck Assessment values will be calculated by descriptive statistics. Mean, standard deviation, and percentiles (1, 5, 10, 25, 50, 75, 90, 95, 99) of the scores will be calculated for each individual assessment.

SECONDARY OUTCOMES:
Test-retest reliability of BrainCheck Assessment values between two different time points | 5 months
  Evaluate the test-retest reliability of BrainCheck assessments using Pearson Correlation coefficients on the descriptive statistics of each individual assessment.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - BrainCheck, Palo Alto, California
  - Maplewood Senior Living, Multiple Locations, Connecticut
  - BrainCheck, Austin, Texas
  - BrainCheck, Houston, Texas
  - BrainCheck, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No